CLINICAL TRIAL: NCT02713893
Title: A Phase I Study of a Novel Intravaginal Antimycotic Cream (Econazole Nitrate 1% Plus Benzydamine HCl 0.12%) Administered Once Daily for 15 Days to Healthy Women
Brief Title: Tolerability and Pharmacokinetic Study of Econazole Nitrate and Benzydamine HCl Intravaginal Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 030(4A)HO14387; CRO-PK-14-289 (Other: CROSS Research S.A., Phase I Unit)
Record Dates: First submitted 2015-08-07; First posted 2016-03-21 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Econazole nitrate 1%; Benzydamine HCl 0.12%; Intravaginal cream; Antimycotic; Tolerability
MeSH Terms: interventions — Econazole; Benzydamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Econazole nitrate 1% plus Benzydamine HCl 0.12% (Experimental): 5 grams of Econazole nitrate 1% plus Benzydamine HCl 0.12% intravaginal cream, once daily for 15 consecutive days
  Interventions: Drug: Econazole nitrate 1% plus Benzydamine HCl 0.12% intravaginal cream
- Placebo plus Econazole nitrate 1% (Active Comparator): 5 grams of Placebo plus Econazole nitrate 1% intravaginal cream, once daily for 15 consecutive days
  Interventions: Drug: Placebo plus Econazole nitrate 1% intravaginal cream
- Placebo plus Benzydamine HCl 0.12% (Active Comparator): 5 grams of Placebo plus Benzydamine HCl 0.12% intravaginal cream, once daily for 15 consecutive days.
  Interventions: Drug: Placebo plus Benzydamine HCl 0.12% intravaginal cream
- Placebo (Placebo Comparator): 5 grams of Placebo intravaginal cream, once daily for 15 consecutive days.
  Interventions: Drug: Placebo intravaginal cream

INTERVENTIONS:
Drug: Econazole nitrate 1% plus Benzydamine HCl 0.12% intravaginal cream
  Arms: Econazole nitrate 1% plus Benzydamine HCl 0.12%
Drug: Placebo plus Econazole nitrate 1% intravaginal cream
  Arms: Placebo plus Econazole nitrate 1%
Drug: Placebo plus Benzydamine HCl 0.12% intravaginal cream
  Arms: Placebo plus Benzydamine HCl 0.12%
Drug: Placebo intravaginal cream
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate local tolerability of the new Econazole/Benzydamine product, in comparison with the Econazole and Benzydamine stand-alone products and placebo. Pharmacokinetics of the study products after single and repeated applications once a day for 15 days, safety of the investigational products and comfort of use will also be evaluated as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study;
2. Sex and age: females, aged 18-55 years old inclusive;
3. Body Mass Index (BMI): 18.5-30 kg/m2 inclusive;
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest (sitting position);
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study;
6. Sexual abstinence: agreement to sexual abstinence during the study;
7. Contraception and fertility: women of child-bearing potential, even if sexual abstinent during the study as required by the study inclusion criteria, must be using at least one reliable method of contraception, as follows:

   1. hormonal oral, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit;
   2. a non-hormonal intrauterine device [IUD] for at least 2 months before the screening visit;
   3. a male sexual partner who agrees to use a male condom;
   4. a vasectomised sexual partner. Female participants of non-child-bearing potential will be admitted. For all female subjects, pregnancy test result must be negative at screening and at each scheduled evaluation;
8. PAP test: negative result at PAP test (i.e. normal PAP test result without atypical cells) at screening.

Exclusion Criteria:

1. ECG (12-leads, supine position): clinically significant abnormalities;
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study as judged by the investigator;
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness;
4. Allergy: ascertained or presumptive hypersensitivity (including allergies) to the active ingredients (econazole and/ or benzydamine) and/or formulations' excipients or related drugs, e.g. other azoles; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study;
5. Diseases: relevant history of renal, hepatic, gastrointestinal, genitourinary, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study or affect the subject's safety;
6. Genitourinary disease: presence of any specific genitourinary symptoms detected at Visit 2 with the relevant questionnaire (genitourinary symptoms questionnaire);
7. Infection history: history of bacterial urinary tract or bacterial and fungal vaginal infections for 3 weeks before the screening visit;
8. Infections: bacterial or fungal infections (microbiology assessment);
9. Gynaecological findings: clinically significant abnormal findings at the gynaecological visit performed by the study gynaecologist;
10. Mucosa conditions: altered mucosa conditions affecting the site of application (e.g. open lesion or other);
11. Vaginal conditions: use of vaginal detergents, soaps and washes that, in the investigator's opinion, may have an influence on vaginal pH and/or change the vaginal flora;
12. Medications: any medication (topical or systemic), including over the counter, herbal medication, topical drugs on the application area and anticoagulants, such as warfarin and acenocoumarol, for 2 weeks before the start of the study. Hormonal contraceptives and hormonal replacement therapies are allowed. Paracetamol will be allowed as a counter-measure for adverse events, on a case by case basis, if deemed appropriate by the investigator;
13. Investigative drug studies: participation in the evaluation of any drug for 3 months before this study, calculated from the first day of the month following the last visit of a previous study and the first day of the present study (date of the informed consent signature);
14. Blood donation: blood donations for 3 months before this study;
15. Drug, alcohol, caffeine, tobacco: history of drug, alcohol (> 1 drink/day, defined according to USDA Dietary Guidelines 2010), tobacco (≥ 10 cigarettes/day) or caffeine (> 5 cups coffee/tea/day) abuse;
16. Diet: Abnormal diets (< 1600 or > 3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
17. Pregnancy: positive or missing pregnancy test at screening or day 1, pregnant or lactating women or females of child-bearing potential not following adequate contraceptive procedures;
18. Non-compliance: subjects suspected to have a high potential for non-compliance to the study procedures according to the investigator's judgement, including non-compliance to sexual abstinence during the study;
19. Drug test (cocaine, amphetamine, methamphetamine, cannabinoids, opiates and ecstasy): positive result at the drug test at screening
20. Alcohol test: positive alcohol breath test at day 1

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Local Adverse Events (AEs) | Up to 7 days after administration
  Occurrence of local Adverse Events (AEs) reported in the subject's diary as 1-3 scores for pruritus, burning sensation, pain, stinging, dryness; occurrence of all the other local AEs referred by the subject; occurrence of all the local Adverse Drug Reactions (ADRs) revealed by the Investigator

SECONDARY OUTCOMES:
Econazole (free base), benzydamine (free base) and benzydamine N-oxide (free base) plasma concentrations | At pre-dose (0), 1, 2, 3, 4, 6, 8, 12, 24 hours after the first (days 1-2) and the last dose (days 15-16) and at pre-dose (0) on day 6±1, day 9±1 and day 12±1
Area under the plasma concentration versus time curve [AUC(0-t)] of econazole (free base), benzydamine (free base) and benzydamine N-oxide (free base) | At pre-dose (0), 1, 2, 3, 4, 6, 8, 12, 24 hours after the first (days 1-2) and the last dose (days 15-16) and at pre-dose (0) on day 6±1, day 9±1 and day 12±1
Treatment Emergent Adverse Events (TEAEs) | 15-16 days
Change from screening in vital signs | From screening (from day -21 to day -7) at days 1 and 15 at pre-dose (0), 12 and 24 hours post-dose
Change from screening in 12-leads ECG | From screening (from day -21 to day -7) at final visit (from day 17 to day 20)
Change from screening in laboratory parameters | From screening (from day -21 to day -7) and at final visit (from day 17 to day 20)
Change from screening in vaginal pH measurement | From screening (from day -21 to day -7), before the application on days 1, 2, 15, on days 6±1, 9±1, 12±1 at final visit (from day 17 to day 20)
Change from screening in gynaecological examination findings | From screening (from day -21 to day -7) at final visit (from day 17 to day 20)
Overall tolerability assessment scale | At final visit (from day 17 to day 20)
Questionnaire for the comfort of use | At final visit (from day 17 to day 20)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — Cross Research S.A.
Locations (1):
- CROSS Research S.A., Phase I Unit, Arzo, Switzerland

IPD SHARING:
Plan to Share IPD: No